CLINICAL TRIAL: NCT02730364
Title: An Open-label, Multicenter, Randomized, Parallel Group, Single-dose Study to Assess the Short Term Efficacy and Safety of Paracetamol 500 mg + Phenylephrine HCl 10 mg + Pheniramine Maleate 20 mg + Vitamin C 200 mg Powder for Oral Solution in Subjects With Symptoms of an Upper Respiratory Tract Infection
Brief Title: An Efficacy and Safety Study of Theraflu Night Powder as Oral Solution for Cold and Flu
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The clinical phase of the study (from FSFV to LSLV) was never initiated due to the sponsor's decision.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205637
Record Dates: First submitted 2016-02-01; First posted 2016-04-06 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Infections, Respiratory Tract
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Acetaminophen; Oxymetazoline; Pheniramine; Ascorbic Acid; Solutions

STUDY DESIGN:
Masking Description: This was an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theraflu night powder (Experimental): Participants will receive a single dose (1 sachet) of Theraflu Night powder containing paracetamol, phenylephrine HCl, pheniramine maleate, and vitamin C as oral solution.
  Interventions: Drug: Paracetamol, phenylephrine HCl, pheniramine maleate, and vitamin C
- No Treatment (No Intervention): Participants in this arm will not receive any medication

INTERVENTIONS:
Drug: Paracetamol, phenylephrine HCl, pheniramine maleate, and vitamin C — One sachet is provided for each participant randomized to the Theraflu Night powder containing paracetamol, phenylephrine HCl, pheniramine maleate, and vitamin C as oral solution.
  Other Names: Theraflu Night powder for oral solution
  Arms: Theraflu night powder

SUMMARY:
The purpose of the study is to assess the short term efficacy of the Theraflu Night powder for oral solution in the Russian population in "Short term relief of the symptoms of colds, chills and influenza, including mild to moderate pain, fever and nasal congestion".

ELIGIBILITY:
Inclusion Criteria:

* Participants must understand and provide written informed consent before any assessment is performed, understand the study procedures, and be willing and able to complete the required assessments
* Males and females ≥ 18 years
* Clinical diagnosis of a URTI as diagnosed by the investigator
* Mild to moderate sore throat, i.e. rated as 1 or 2 on a 4-point ordinal scale (0=not present, 1= mild, 2=moderate, 3=severe), or headache (1, 2 or 3) or fever (less than 39°C ) or/and Nasal congestion (blocked nose): may be accompanied by rhinorrhea (runny nose) and/or sneezing
* Baseline Jackson TSS > 8
* Common cold symptoms for less than 48 hours

Exclusion Criteria:

* Use of other investigational drugs within 30 days or 5 half-lives of enrollment, whichever is longer. Investigational drug refers to any drug being evaluated in clinical trials
* History of or known hypersensitivity to any of the study drugs, excipients or to drugs of similar chemical classes
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL) or urine dipstick at baseline
* Any history of drug hypersensitivity, asthma, urticaria, or other significant allergic diathesis. Participants with uncomplicated seasonal allergic rhinitis can be accepted if expected allergy season is clearly one month outside enrollment/ treatment period
* Any history of brain diseases, liver diseases or epilepsy
* Any evidence of uncontrolled cardiovascular (including hypertension), pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinological, metabolic, neurological or psychiatric diseases at screening
* Subject has closed angle glaucoma, urinary retention, prostatic hyperplasia, pyloroduodenal obstruction, pheochromocytoma, diabetes mellitus
* A positive alcohol breath test or positive urine drug screen or a medical history data indicative of alcoholism, drug addiction, or drug abuse within the preceding 2 years
* Subject is current smoker of ≥10 cigarettes per day (or reports equivalent smoking habits using other tobacco products) and is unwilling to refrain from smoking while at the study site
* Subject is current smoker of ≥10 cigarettes per day (or reports equivalent smoking habits using other tobacco products) and is unwilling to refrain from smoking while at the study site
* Subject is taking or has taken within the last two weeks of dosing monoamine oxidase inhibitors, antidepressants, atropine, beta-blocking or sympathomimetic drugs desferrioxamine, hepatotoxic drugs, drugs inducing liver microsomal enzyme, (such as phenytoin, carbamazepine, isoniazid and rifampicin), neuroleptic drugs, chlorzoxazone, CNS depressant drugs including barbiturates, hypnotics, opioid analgesics, anxiolytic sedatives, antipsychotics or is anticipated to require any of these medications at any time throughout the study
* Subject has used: Systemic or topical corticosteroids (with the exception of HRT and contraceptive steroids for females), within 3 weeks prior to dosing or Slow-release steroids (with the exception of HRT and contraceptive steroids for females) within 90 days prior to dosing
* Subject has used any of the following medications within 6 hours before first study drug administration, or is anticipated to use any of these medications at any time throughout the study: Any inhaler, medicated confectionary, throat lozenges, throat pastilles, sprays, any products with demulcent properties such as chewing gums and boiled sweets or mints, Any medication for sore throat containing a local anaesthetic, Cold products and oral nasal decongestant products, Paracetamol or any NSAID
* Subject has used substances of abuse, herbal medicines, antihistamines and homeopathic medicine within 72 hours of dosing or is anticipated to require any of these drugs at any time throughout the study
* Subject was previously enrolled into the current study
* Persons directly or indirectly involved in the execution of this protocol, including first degree relative of a study investigator, employees of the clinical study site, employees of the CRO and persons related to them
* "Vulnerable" individual (as defined by the IRB e.g. incarcerated person)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Estimated); Primary Completion 2017-04-01 (Estimated); Study Completion 2017-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy assessment Change from baseline, 3 hours after dosing in the Jackson Total Symptom Score (JTSS) | At 3 hours post dosing
  The severity of common cold symptoms will be self-assessed using the Jackson 8 items scale (questionnaire) by the participants on the site. This questionnaire measures the severity of 5 local symptoms (nasal congestion, rhinorrhea, sneezing, cough, and sore throat) and 3 systemic symptoms (chilliness, headache, malaise) each on a 4-point ordinal scale (0=not present, 1= mild, 2=moderate, 3= severe).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline